CLINICAL TRIAL: NCT05646329
Title: The Effect Of Online Individual Motivational Interviewing Applied To Nursing Students On Problematic Internet Use And Loneliness Level
Brief Title: The Effect of Motivational Interviewing on Problematic Internet Use and Loneliness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Elif Altun, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Elif Altun
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Problematic Internet Use; Loneliness
Keywords: Motivational Interviewing; Problematic Internet Use; University students; Psychosocial Intervention; Loneliness
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: In the study, 66 students were taken as sampling, 33 of which were experimental and 33 were control.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, it was not possible to blind the researcher and the participant who applied the intervention, but the statistics and report writing process were blinded.The students in the experimental and control groups related to the research were informed about the purpose of the study.The person conducting the research knows which is the experimental group and which is the control group. For this reason, single and double blinding was not done in the study. The data regarding the measurements were written as 'A' and 'B' without specifying the experimental and control groups, and the groups were coded.The analysis of the data coded in terms of groups will be done by the statistics expert. After the statistical analyzes are made and the research report is written, the coding for the experimental and control groups will be explained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The motivational interview to be held with the experimental group was planned as 4 sessions together with the follow-up session. The session will last a maximum of 40 minutes. The session will be once a week. Motivational interview will be conducted individually and online with the experimental group. For individual interviews, the appropriate day and time will be determined with the researcher before the first session and the sessions will continue on the same day and time every week.
  Interventions: Behavioral: Motivational Interview
- Waiting list group (No Intervention): If the students in the control group make a request at the end of the study, an online individual motivational interview will be held. The intervention applied to the experimental group will also be applied to the control group at the end of the study.
  Intervention: Behavioural Intervention Based on Problematic Internet Use

INTERVENTIONS:
Behavioral: Motivational Interview — The motivational interview to be held with the experimental group was planned as 4 sessions together with the follow-up session.
  Arms: Experimental

SUMMARY:
This research will examine the effect of online individual motivational interviewing applied to nursing students on problematic internet use and loneliness. Mixed method will be used in the research.

DETAILED DESCRIPTION:
Problematic internet use is seen as a multidimensional syndrome consisting of cognitive and behavioral symptoms that cause negative social, academic and professional consequences. Problematic internet use to the individual; psychological effects such as eating disorder, depression, sleep disorder, addiction, anxiety, physical effects such as injury, posture disorders, social effects such as lack of social relations and loneliness. Many issues related to problematic internet use are mentioned. However, psychosocial intervention studies to help problematic internet use remain a subject of little research.

ELIGIBILITY:
Inclusion Criteria:

1. Being in the pre-intention or intention stage according to the motivational interview change cycle determination form,
2. Scoring above the problematic internet use scale average,
3. Volunteer to participate in the study,
4. Having no problems with speaking and understanding Turkish

Exclusion Criteria:

1. Having a psychiatric diagnosis
2. Receiving ongoing individual or group counseling
3. Being in the phase of preparation, action or maintenance from the change phases
4. Not wanting to continue research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Change of Problematic Internet Use | baseline, week 3 , 3- month follow up (Pretest-posttest follow-up experimental design)]
  The 33-item Problematic Internet Use Scale will measure the severity of problematic internet use. Problematic Internet Use Scale is measure designed to assess the symptoms of problematic internet use, with a higher total score suggesting more severe problematic use symptoms. Scores range from 33 to 165.

SECONDARY OUTCOMES:
Change of Social and Emotional Loneliness Scale for Adults | baseline, week 3 , 3- month follow up (Pretest-posttest follow-up experimental design)
  The 15-item Social and Emotional Loneliness Scale for Adults will measure the severity of social and emotional loneliness. Social and Emotional Loneliness Scale for Adults is measure designed to assess the symptoms of social and emotional loneliness, with a higher total score suggesting more severe social and emotional loneliness. Scores range from 15 to 105.

OTHER OUTCOMES:
Participant information form | baseline
  Participant information form; It consists of 6 questions prepared by the researcher to determine the sociodemographic characteristics of the student participating in the research
Change of Motivational Interview Change Cycle Determination Form | baseline, week 3, 3-month follow up
  Motivational Interview Change Cycle Determination Form It is the form that will be used in the research to determine the place in the Change Cycle before being included in the motivational interview, and to determine what stage they are in after the interview. The form consists of 14 questions and was created by the researcher.
Online Individual Motivational Interview Evaluation Form-Student | 3-month follow up
  Online Individual Motivational Interview Evaluation Form-Student It was prepared by the researcher in order to reveal the opinions of the students participating in the motivational interview on the evaluation of motivational interviewing, and it is a form containing 7 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Altun, Principal Investigator — elifaltun@gazi.edu.tr
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: July 2023- Novamber 2023

REFERENCES:
- [Result] Guo L, Luo M, Wang WX, Huang GL, Xu Y, Gao X, Lu CY, Zhang WH. Association between problematic Internet use, sleep disturbance, and suicidal behavior in Chinese adolescents. J Behav Addict. 2018 Dec 1;7(4):965-975. doi: 10.1556/2006.7.2018.115. Epub 2018 Nov 26. PMID 30474380
- [Result] Odacı, H. ve Kalkan, M. (2010). Problematic Internet use, loneliness and dating anxiety among young adult university students. Computers & Education, 55(3), 1091-1097.
- [Result] Park S, Hong KE, Park EJ, Ha KS, Yoo HJ. The association between problematic internet use and depression, suicidal ideation and bipolar disorder symptoms in Korean adolescents. Aust N Z J Psychiatry. 2013 Feb;47(2):153-9. doi: 10.1177/0004867412463613. Epub 2012 Oct 9. PMID 23047959
- [Result] Shek, D. T., Sun, R. C., and Yu, L. (2013). Internet addiction. Springer.
- [Result] Tao ZL, Liu Y. Is there a relationship between Internet dependence and eating disorders? A comparison study of Internet dependents and non-Internet dependents. Eat Weight Disord. 2009 Jun-Sep;14(2-3):e77-83. doi: 10.1007/BF03327803. PMID 19934640
- [Result] Kim HJ, Min JY, Kim HJ, Min KB. Accident risk associated with smartphone addiction: A study on university students in Korea. J Behav Addict. 2017 Dec 1;6(4):699-707. doi: 10.1556/2006.6.2017.070. Epub 2017 Nov 3. PMID 29099234
- [Result] Makhsous M, Lin F, Hendrix RW, Hepler M, Zhang LQ. Sitting with adjustable ischial and back supports: biomechanical changes. Spine (Phila Pa 1976). 2003 Jun 1;28(11):1113-21; discussion 1121-2. doi: 10.1097/01.BRS.0000068243.63203.A8. PMID 12782977